CLINICAL TRIAL: NCT05222815
Title: Comparing Fingerstick Blood Glucose Monitoring Versus Continuous Glucose Monitoring in Primary Care
Brief Title: Glucose Monitoring Comparison in Primary Care
Acronym: GluCoCare
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-326
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; Continuous Glucose Monitor; Blood Glucose Monitor; Self-Monitoring of Blood Glucose; Primary Care; Glycemic Control; Time In Range; Diabetes Distress; Insulin; A1C; Glucose Management; Comparative effectiveness
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGM (continuous glucose monitoring) (Experimental): Use CGM, with availability of Ambulatory Glucose Profile (AGP) data, to monitor and manage glucose over 12 months, in individuals with type 2 diabetes on insulin with or without other glycemic therapies. Glucose management over the 12 months study period will be in primary care, using "usual care" resources.
  Interventions: Other: CGM
- SMBG (Self-monitoring of blood glucose) (Active Comparator): Use SMBG, as currently used in primary care, to monitor and manage glucose over 12 months, in individuals with type 2 diabetes on insulin with or without other glycemic therapies. Glucose management over the 12 months study period will be in primary care, using "usual care" resources.
  Interventions: Other: SMBG

INTERVENTIONS:
Other: CGM — Continuous glucose monitor (CGM)-based glucose monitoring
  Arms: CGM (continuous glucose monitoring)
Other: SMBG — Self-monitoring of blood glucose (SMBG)-based glucose monitoring
  Arms: SMBG (Self-monitoring of blood glucose)

SUMMARY:
This research trial will randomize 50 primary care clinics and 354 patients in accordance with their primary care clinic assignment to 2 different glucose monitoring strategies (SMBG vs. CGM) and compare the effectiveness through a pragmatic clinic cluster randomized design, with active glycemic management in a "usual" primary care setting, over the course of a 12 month active study period.

DETAILED DESCRIPTION:
The trial will evaluate the comparative effectiveness of SMBG (self-monitoring of blood glucose, also known as blood glucose monitoring [BGM] or fingerstick blood glucose monitoring) vs. continuous glucose monitoring (CGM), in managing glucose levels in individuals with type 2 diabetes (T2D) using insulin, with or without other glycemic therapies, in a primary care setting.

The study will use a 2-arm, parallel group, cluster-randomized trial over a 12-month period. 50 primary care clinics will be randomly assigned to either use SMBG for glucose monitoring (25 clinics), with ongoing glycemic management provided by usual care in primary care, or CGM for glucose monitoring (25 clinics), with ongoing glycemic management provided by usual care in primary care using CGM and Ambulatory Glucose Profile (AGP) reports in a typical clinic setting. The study will use glycemic monitoring devices available to participants using real-world resources to cover the cost of the devices, and will be fundamentally pragmatic in nature.

354 patients (approximately 7/clinic) will be enrolled over 13 months (12 months of active intervention) with an intention-to-treat primary analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 (inclusive)
2. Diagnosis of type 2 diabetes
3. A1C 7.5% to 12% (inclusive) in the last 2 months. (If A1C is older than 2 months at the baseline visit, a point-of-care or lab A1C may be done for eligibility)
4. Insulin use with or without other classes of glycemia medication use
5. No significant comorbidities that could impair the ability of a primary care team to manage diabetes, including but not limited to end stage renal disease, cognitive impairment, active cancer, and pregnancy
6. Established care within the HealthPartners Care Group, no plans to move within the next year, and willing to participate for the duration of the study
7. Willing and able to follow procedures for collecting blinded CGM data at baseline, 6 and 12 months follow-up
8. Willing to complete surveys at baseline, 3, 6, 9 and 12 months.
9. Willing to use SMBG or CGM, depending on randomization, in the way that their care team recommends and/or how they feel is most useful in managing their diabetes
10. Not currently using personal CGM
11. Not planning to become pregnant

Exclusion Criteria:

1. Unwillingness or inability to provide informed consent
2. Deemed not suitable for participation in the study based on any other clinical criteria as determined by study investigator(s)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in A1C | 12 months
  To evaluate the effectiveness of two glucose monitoring strategies to reduce A1C levels by measuring differential within-patient change by study arm in A1C (%) from baseline to 12 months.
Change in Diabetes Distress | 12 months
  To evaluate the effectiveness of two glucose monitoring strategies to reduce diabetes distress by measuring differential within-patient change by study arm in Diabetes Distress Scale scores from baseline to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Bergenstal, MD, Principal Investigator — International Diabetes Center, HealthPartners Institute; Thomas W Martens, MD, Principal Investigator — International Diabetes Center, HealthPartners Institute
Locations (1):
- International Diabetes Center, Saint Louis Park, Minnesota, United States